CLINICAL TRIAL: NCT05932524
Title: Low-dose Baricitinib Plus High-dose Dexamethasone as First-line Treatment for Patients With Newly Diagnosed Immune Thrombocytopenia: a Multicenter, Open-label, Randomized, Controlled, Phase 2 Trial
Brief Title: Low-dose Baricitinib Plus High-dose Dexamethasone for Patients With Newly Diagnosed Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Luhe Hospital (Other); Chinese PLA General Hospital (Other); Navy General Hospital, Beijing (Other); Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-BAITP-03
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Immune Thrombocytopenia
Keywords: Baricitinib; High-dose dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — baricitinib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned at a 1:1 ratio to receive baricitinib plus high-dose dexamethasone or high-dose dexamethasone alone. Each group requires 66 patients (considering 10% drop-off).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose baricitinib plus high-dose dexamethasone (Experimental): Oral baricitinib is given at a dose of 2 mg daily for 6 consecutive months. Dexamethasone is administrated at 40 mg per day for 4 consecutive days (the 4-day course of dexamethasone will be repeated in the case of lack of response by day 10). Treatment will be discontinued if very severe or life-threatening adverse events developed or at the patients' request.
  Interventions: Drug: Baricitinib 2 MG; Drug: Dexamethasone
- High-dose dexamethasone (Active Comparator): Dexamethasone is administrated at 40 mg per day for 4 consecutive days (the 4-day course of dexamethasone will be repeated in the case of lack of response by day 10). Treatment will be discontinued if very severe or life-threatening adverse events developed or at the patients' request.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Baricitinib 2 MG — Baricitinib 2 mg q.d., p.o., for 6 consecutive months.
  Other Names: Olumiant
  Arms: Low-dose baricitinib plus high-dose dexamethasone
Drug: Dexamethasone — Dexamethasone 40 mg q.d. for 4 consecutive days (the 4-day course of dexamethasone will be repeated in the case of lack of response by day 10)
  Other Names: HD-DXM

SUMMARY:
A randomized, open-label, multicenter, phase 2 trial to compare the efficacy and safety of baricitinib plus high-dose dexamethasone compared to high-dose dexamethasone monotherapy for the first-line treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This is a parallel group, multicenter, randomized, controlled trial of patients with ITP in China. Patients were randomly assigned to receive baricitinib plus high-dose dexamethasone or high-dose dexamethasone monotherapy. Treatment will be discontinued if very severe or life-threatening adverse events developed or at the patients' request. The primary endpoint is durable response, defined as the maintenance of platelet count ≥30,000/μL and at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed newly-diagnosed, treatment-naive ITP;
2. A platelet count <30,000/μL, or a platelet count <50,000/μL with clinically significant bleeding symptoms (WHO bleeding scale 2 or above) at the enrollment;
3. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
2. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
3. Active or a history of malignancy;
4. Pregnancy or lactation;
5. Received first-line and second-line ITP-modifying therapy;
6. Previously received corticosteroids or immunosuppressive agents for non-ITP diseases within 6 months before enrollment;
7. A history of clinically significant adverse reactions to previous corticosteroid therapy;
8. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia);
9. Current or recent (<4 weeks prior to screening) clinically serious viral, bacterial, fungal, or parasitic infection;
10. A history of symptomatic herpes zoster infection within 12 weeks prior to screening;
11. Active or chronic viral infection from hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV);
12. Have evidence of active tuberculosis (TB), or have previously had evidence of active TB and did not receive appropriate and documented treatment, or have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB;
13. Have experienced a clinically significant thrombotic event within 24 weeks of screening or are on anticoagulants and in the opinion of the investigator are not well controlled;
14. Myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure;
15. A history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data;
16. Any of the following specific abnormalities on screening laboratory tests:

1) ALT or AST >2 x ULN, or total bilirubin ≥1.5 x ULN 2) hemoglobin <9 g/dL, or total white blood cell (WBC) count <2,500/µL, or neutropenia (absolute neutrophil count <1,200/µL), or lymphopenia (lymphocyte count <750/µL) 3) eGFR <50 mL/min/1.73 m^2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Durable response | 6 months
  The maintenance of a platelet count ≥30,000/μL, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Complete response (CR) | 1 month
  A platelet count over 100,000/μL and absence of bleeding.
Response (R) | 1 month
  A platelet count over 30,000/μL and at least 2-fold increase of the baseline count and absence of bleeding.
Time to response | 6 months
  The time from starting treatment to time of achievement of CR or R.
Duration of response | 6 months
  Duration of response at 6-month follow up.
Early response | 7 days
  Achievement of CR or R at day 7
Initial response | 28 days
  Achievement of CR or R at day 28
Bleeding events | From the start of study treatment (Day 1) to the end of week 26
  Clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale.
Health-related quality of life (HRQoL) | From the start of study treatment (Day 1) to the end of week 26
  ITP-PAQ is used to assess the Health Related Quality of Life (HRQoL) before and after treatment.
Adverse events | From the start of study treatment (Day 1) to the end of week 26
  Adverse events (AEs) are reported and graded in accordance with the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (10):
- China (10):
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Beijing Tsinghua Changgeng Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Sixth Medical Center of PLA General Hospital, Beijing